CLINICAL TRIAL: NCT03064230
Title: Promotion and Protection of the Well Being of Women Athletes Through the Female Athlete Triad Screening
Brief Title: Promotion of Wellbeing in Women Athletes
Acronym: Wsport
Status: Completed | Type: Observational
Sponsor: Campus Bio-Medico University (Other)
Collaborators: Federazione medicina sportiva italiana (FMSI) (Unknown)
Responsible Party: Principal Investigator, Roberto Angioli, Professor, Campus Bio-Medico University
Other Study IDs: 25/15 OSS ComEt CBM
Record Dates: First submitted 2017-02-19; First posted 2017-02-27 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Quality of Life

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Athletes agonists (Experimental Group): I) age between 14 and 40 years who met the definition of competitive sports athletes adopted by the Italian Ministry of Health II) absence of malignancies; III) informed consent obtained from the patient; IV) no previous surgical, chemotherapic and/or radiotherapic treatments.
  We excluded all patients who presented any conditions that could alter quality of life such as: I) recent traumas; II) recent surgeries; III) oncologic history; IV) uncontrolled systemic illnesses; V) severe or uncontrolled infection; VI) mental illness; VII) pregnancy.
  QoL questionnaire SF-12 and and a screening questionnaire were requested
  Interventions: Other: QoL questionnaire SF-12 and and a screening questionnaire
- women not agonists (Control Group): I) age between 14 and 40 years who did not met the definition of competitive sports athletes adopted by the Italian Ministry of Health; II) absence of malignancies; III) informed consent obtained from the patient; IV) no previous surgical, chemotherapic and/or radiotherapic treatments.
  We excluded all patients who presented any conditions that could alter quality of life such as: I) recent traumas; II) recent surgeries; III) oncologic history; IV) uncontrolled systemic illnesses; V) severe or uncontrolled infection; VI) mental illness; VII) pregnancy. QoL questionnaire SF-12 and and a screening questionnaire were requested
  Interventions: Other: QoL questionnaire SF-12 and and a screening questionnaire

INTERVENTIONS:
Other: QoL questionnaire SF-12 and and a screening questionnaire — patient were asked to fill questionnaires

SUMMARY:
The Female Athlete Triad is a medical condition often observed in physically active girls and women, and involves 3 components: (1) low energy availability with or without disordered eating, (2) menstrual dysfunction, and (3) low bone mineral density. An early intervention is essential to prevent its progression to serious endpoints including clinical eating disorders, amenorrhea, and osteoporosis that can affect the quality of life of these patients and even compromise the athletic performance.

All patients, aged between 14 and 40 years, who met the inclusion and exclusion criteria, were prospectively enrolled in this observational study and were divided into two groups: Athletes agonists (Experimental Group or Group A) and women who do not perform agonistic sports (Control Group or Group B). In both groups of patients, the investigators administered two types of questionnaires: a standardized quality of Life questionnaire, validated in Italian (SF-12) and a screening questionnaire recommended by the Female Athlete Triad Expert Panel.

DETAILED DESCRIPTION:
From January 2016 to May 2016 the investigators considered eligible all consecutive women, aged between 14 and 40 years, who came to undergo routine physical examination.

The institutional internal review board approved the study. Inclusion criteria were: I) age between 14 and 40 years; II) absence of malignancies; III) informed consent obtained from the patient; IV) no previous surgical, chemotherapic and/or radiotherapic treatments.

the investigators excluded all patients who presented any conditions that could alter quality of life such as: I) recent traumas; II) recent surgeries; III) oncologic history; IV) uncontrolled systemic illnesses; V) severe or uncontrolled infection; VI) mental illness; VII) pregnancy.

All patients who met the inclusion and exclusion criteria were prospectively enrolled in this observational study and were divided into two groups: Athletes agonists (Experimental Group or Group A) and women who do not perform any agonistic sports (Control Group or Group B).

Were considered agonists athletes and enrolled in Group A all the patients who met the definition of competitive sports athletes adopted by the Italian Ministry of Health (Ministerial Decree, D.M. 18/02/1982 - Circular No. 7 of 01/31/1983): "form of sporting activity systematically and/or continually practiced, especially organized by the National Sports Federations, the Sporting Promotion bodies recognized both by CONI and the Ministry of Education with regard to the Youth Games at National level, to the achievement of a certain level of sportive performance". All other women were considered as not athletes and were included in the control group (Group B).

To assess the sample size, in order to detect a difference of 3 points in SF12-questionnaires, were used the Cohen formulas, considering a power of 80% (two-tails; P = 0.05 Long Rank Test): 100 patients were necessary for each group to detect a statistically significant difference.

In all patients an accurate gynecological history was recorded with a special focus on menstrual irregularities, from the age of menarche to present. It was also investigated the presence of other gynecological symptoms that can affect athletic performance of the patient, such as pain during menstruation (dysmenorrhea) or other forms of pelvic pain.

A registration of medication history was taken, including medications that can affect menstruation and /or bone mass density (BMD), as contraceptive pills or other contraceptive agents.

Moreover all patients underwent the evaluation of every physical characteristics that could be suggestive of an eating disorders, such as low body mass index (BMI), weight loss, orthostatic hypotension, swelling of the parotid glands or presence of calluses on the proximal interphalangeal joints (also known as Mark Russell). Finally an accurate record of all the previous episodes of bone stress, injuries and fractures was recorded.

In both groups of patients two types of questionnaires were administrated: a standardized quality of Life questionnaire, validated in Italian (SF-12) and a screening questionnaire (the same that the Female Athlete Triad Expert Panel recommends as a screening and an integral part of the athletes routine physical assessment) aimed to the identification of apparatus-specific dysfunctions (Female Athlete Triad). Even if this last questionnaire is still not validated in Italian, both questionnaires (SF-12 and screening) were administered in Italian.

SF-12 questionnaire is considered a reliable measure of perceived health that describes the degree of general physical health status and mental health distress. It consists of 12 items, derived from the physical and mental domains. SF-12 was considered altered if the score was <40, either from the physical or mental functioning point of view, because means of 50 and standard deviations of 10 are usually achieved in the general population.

The screening questionnaire was focused on those main risk factors that can lead to a decreased quality of life in women and to an early detection of a medical dysfunction related to the female triad. the investigators used two different cut-off to consider the questionnaire altered: 1) alteration of at least two items of the questionnaire; 2) alteration of at least two items of the questionnaire, where question 6,7 and 8 (all related to eating disorders) were considered as one.

If either one of the two questionnaire resulted altered, or would arise any suspicion from the physical evaluation, the patient was sent to a more in-depth assessment in order to verify the presence of a clinical dysfunction.

Finally all the data were recorded in a database. The incidence and prevalence of gynecological disorders were calculated.

Spearman correlation test was used to assess if altered levels of quality of life corresponded to an alteration of the screening questionnaire and if an alteration of the screening questionnaire effectively corresponded, after a more in-depth clinical assessment, to a clinical dysfunction. Correlation coefficients whose magnitude were between 0.9 and 1.0 indicated variables which could be considered very highly correlated. Correlation coefficients whose magnitude were between 0.7 and 0.9 indicated variables which could be considered highly correlated. Correlation coefficients whose magnitude were between 0.5 and 0.7 indicated variables which could be considered moderately correlated. Correlation coefficients whose magnitude were between 0.3 and 0.5 indicated variables which had a low correlation. Correlation coefficients whose magnitude were <0.3 had little if any (linear) correlation.

The sensitivity, specificity, positive (PPV) and negative (NPV) predictive values, and accuracy of the screening questionnaire in assessing the presence of a clinical dysfunction were calculated, using the physical examination as the 'gold standard'. The sensitivity, specificity, positive (PPV) and negative (NPV) predictive values, and accuracy of the screening questionnaire in assessing the presence of an alteration of quality of life were calculated, using SF-12 questionnaire as the 'gold standard'.

All continuous data were expressed as mean and standard deviation. All the variables quantitative were compared using the Student's t test or the Mann-Whitney, depending on their distribution pattern. Qualitative variables were compared using the Chisquare or Fisher tests.

For all statistical comparisons, statistical significance was set at P <0.05. Statistical analysis was performed using software Medcalc © statistical software ver. 12.4.0.0.

ELIGIBILITY:
Inclusion Criteria:

1. age between 14 and 40 years;
2. absence of malignancies;
3. informed consent obtained from the patient;
4. no previous surgical, chemotherapic and/or radiotherapic treatments.

Exclusion Criteria:

1. recent traumas;
2. recent surgeries;
3. oncologic history;
4. uncontrolled systemic illnesses;
5. severe or uncontrolled infection;
6. mental illness;
7. pregnancy.

Ages: 14 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — evaluation of well being in female athletes and evaluation of gynecologic dysfunctions
Study Population: Women aged between 14 and 40 years, who came to undergo routine physical examination.All patients who met the inclusion and exclusion criteria were prospectively enrolled in this observational study and were divided into two groups:Athletes agonists(Experimental Group)and women who do not perform any agonistic sports(Control Group). Were considered agonists athletes all the patients who met the definition of competitive sports athletes adopted by the Italian Ministry of Health:"form of sporting activity systematically and/or continually practiced, especially organized by the National Sports Federations with regard to the Youth Games at National level, to the achievement of a certain level of sportive performance".All other women were included in the control group.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-05-30 (Actual); Study Completion 2016-05-30 (Actual)

PRIMARY OUTCOMES:
Quality of life through a validated in Italian (SF-12) and a screening questionnaire recommended by the Female Athlete Triad Expert Panel. | day 1 at time of the visit. no follow/up
  SF-12 questionnaire is a reliable measure of perceived health that describes the degree of general physical health status and mental health distress. It consists of 12 items, derived from the physical and mental domains. In our study SF-12 was considered altered if the score was <40, either from the physical or mental functioning point of view, because means of 50 and standard deviations of 10 are usually achieved in the general population.
  the athlete triad screening questionnaire was focused on those main risk factors that can lead to a decreased quality of life in women and to an early detection of a medical dysfunction related to the female triad. In our study we evaluated two cut-off to consider the questionnaire altered: 1) alteration of at least two items of the questionnaire; 2) alteration of at least two items of the questionnaire, where question 6,7 and 8 (all related to eating disorders) were considered as one.

SECONDARY OUTCOMES:
correlation between altered screening questionnaire and a clinical dysfunction | day 1 and through completion of work-up, average 1 month.
  If either one of the two questionnaire resulted altered (SF-12 or screening questionnaire), or would arise any suspicion from the physical evaluation, the patient was sent to a more in-depth assessment in order to verify the presence of a clinical dysfunction.
Incidence and prevalence of gynecological disorders in female athletes | day 1 and through completion of work-up, average 1 month.
  We compared our results within the two groups to assess if there were any differences in terms of incidence or prevalence of gynecologic disfunctions

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Angioli, Study Chair — University Campus Bio Medico of Rome

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Joy E, De Souza MJ, Nattiv A, Misra M, Williams NI, Mallinson RJ, Gibbs JC, Olmsted M, Goolsby M, Matheson G, Barrack M, Burke L, Drinkwater B, Lebrun C, Loucks AB, Mountjoy M, Nichols J, Borgen JS. 2014 female athlete triad coalition consensus statement on treatment and return to play of the female athlete triad. Curr Sports Med Rep. 2014 Jul-Aug;13(4):219-32. doi: 10.1249/JSR.0000000000000077. PMID 25014387
- See also: female athlete triad — https://www.ncbi.nlm.nih.gov/pubmed/25014387